CLINICAL TRIAL: NCT01707108
Title: Survival and Success of MIS C1 Implants- a Field Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0113-12-RMB CTIL
Record Dates: First submitted 2012-10-11; First posted 2012-10-16 (Estimated); Results first posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Failure of Osseointegration of Dental Implant
Keywords: dental implants; bone loss
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dental Implants (Experimental): Rehabilitation of missing teeth with Dental Implant (MIS Technologies)
  Interventions: Device: Dental Implant (MIS Technologies)

INTERVENTIONS:
Device: Dental Implant (MIS Technologies) — MIS Technologies Ltd. C1 Dental implants

SUMMARY:
The aim of the present study is to evaluate the 1-year and 3-year survival and success of MIS® C1 implants with a length of 10-15mm.

Specific Aims

1. To study 1-year and 3-year implant survival rate C1 implants
2. To study 1-year and 3-year implant bone level changes of C1 implants

DETAILED DESCRIPTION:
10 implants will be allocated to each of the twelve dentists, for a total of 120 implants. One test implant per patient will be allowed into the study for a total of 120 patients.

The following data will be collected for each patient/implant:

1. Patient data including birthdate, health, surgery date.
2. Implant length, diameter
3. Insertion torque
4. Periapical radiographs (at insertion, and twelve months post surgery).
5. Post operative complications and adverse events.
6. Periodontal data around Ramfjord teeth (16, 21, 24, 36, 41, 44) : Plaque index, Gingival Index, Probing depth in six sites and Bleeding on probing in six sites, at baseline and twelve months post surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-75.
2. Patient expresses his wish to restore the missing tooth/teeth with implant therapy.
3. Partial edentulism with available bone height for dental implants ≥ 10mm mm.

Exclusion Criteria:

1. Contraindicating medical conditions such as uncontrolled diabetes, untreated malignancies, pregnancy, previous/current bisphosphonate therapy.
2. Untreated periodontal disease, untreated caries, periapical pathology in contact with the location of the perspective implant.
3. Major bone augmentation in conjunction with implant placement. Localised bone augmentation in conjunction with implant placement, of up to 3 mm on 1-2 aspects of the implant will be allowed.
4. One stage immediate loading/restoration.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-01-28 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Horwitz, DMD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Dental Implants
Groups:
- Dental Implants: Patients with missing teeth that are indicated for rehabilitation with Dental Implants (MIS Technologies) will be recruited. All the implants needed in the surgical area of the recruited patients will be allowed into the study
  Dental Implant (MIS Technologies): MIS Technologies Ltd. C1 Dental implants
Period: Overall Study
Arm/Group | Dental Implants
Started | 60; 117 Dental Implants
1 Year | 60; 117 Dental Implants
Completed | 60; 117 Dental Implants
Not Completed | 0; 0 Dental Implants

BASELINE CHARACTERISTICS:
Units Other Than Participants: implants
Arm/Group | Dental Implants
Number analyzed (Participants) | 60
Number analyzed (implants) | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 47
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  Israel | 60

OUTCOME MEASURES:

1. Primary Outcome: Survival Rate
Description: 1 year survival rate
Time Frame: 1 year post implantation
Population: Fifteen patients (25%) received 1 implant and 45 patients (75%) received 2 or more implants.
Measure: Count of Units; unit: dental implants
Units Other Than Participants: dental implants
Arm/Group | Dental Implants
Number analyzed (Participants) | 60
Number analyzed (dental implants) | 117
dental implants | 115

2. Secondary Outcome: 1 Year Implant Bone Level Changes
Description: bone change in millimeters after 1 year
Time Frame: 1 year post implantation
Population: 117 implants in 60 patients
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: dental implants
Arm/Group | Dental Implants
Number analyzed (Participants) | 60
Number analyzed (dental implants) | 117
millimeters | 0.54 (0.55)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Dental Implants
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-01-24): https://cdn.clinicaltrials.gov/large-docs/08/NCT01707108/Prot_SAP_000.pdf